CLINICAL TRIAL: NCT01373710
Title: Phase 1-2 Study of Safety and Efficacy of Intrathecal Trastuzumab Administration in Metastatic HER2 Positive Breast Cancer Patients Developing Carcinomatous Meningitis
Brief Title: Intrathecal Trastuzumab Administration in Metastatic Breast Cancer Patients Developing Carcinomatous Meningitis
Acronym: HIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Hoffmann-La Roche (Industry); Centre Leon Berard (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Centre Oscar Lambret (Other); Centre Francois Baclesse (Other); Institut Bergonié (Other); University Hospital, Toulouse (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/501/M; 2009-017218-63 (EudraCT Number)
Record Dates: First submitted 2011-05-24; First posted 2011-06-15 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer; Carcinomatous Meningitis
Keywords: Adverse Reaction to Trastuzumab Administered by intrathecal
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab intrathecal (Experimental)
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — One injection per week during 8 weeks by lumbar puncture or Ommaya Reservoir. 4 levels of doses are expected from 30 mg to 150 mg
  Other Names: Herceptin

SUMMARY:
The purpose of this study is:

Phase I: To determine the Trastuzumab maximum tolerated dose (MTD) when weekly administrated by intrathecal or intraventricular route to reach a intra CSF target concentration (30 µg/mL) near the conventional therapeutic concentration and depending on the dose-limiting toxicity (DLT)

Phase II: Determination of antitumor activity trastuzumab when administrated by IT or intra-ventricular in terms of neurological progression-free survival at 2 months

DETAILED DESCRIPTION:
Phase I: Secondary Outcome Measures:

Recommended dose (RD will be used in Phase II) Toxicity during treatment Clinical response to specific neurologic symptoms Time to neurologic progression Biological response: CSF cellularity and protein concentration Radiological response: cerebrospinal meningitis and neuraxis RMI Impact on quality of life Impact on survival (overall survival, survival without neurological progression, progression-free survival) Pharmacokinetics: dose of trastuzumab in CSF and plasma FCGR3A Genetic status influence on efficacy trastuzumab in metastatic breast cancer

Phase II: Secondary Outcome Measures :

Toxicity during treatment Clinical response to specific neurologic symptoms Time to neurologic progression Biological response: CSF cellularity and protein concentration Radiological response: cerebrospinal meningitis and neuraxis MRI Impact on quality of life Impact on survival (overall survival, survival without neurological progression, progression-free survival) Pharmacokinetics: dose of trastuzumab in CSF and plasma (confirmation of phase I data with 5 patients) FCGR3A Genetic status influence on efficacy trastuzumab in metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Metaplastic Infiltrating adenocarcinoma of the breast
* HER2 Overexpression by IHC and / or amplification (FISH and or ICHS)
* Positive diagnosis of neoplastic meningitis: positive CSF cytology (obtained within 28 days before inclusion) AND / OR clinical symptoms of neoplastic meningitis and aspect of tumoral meningitis on MRI
* Brain metastases are allowed without prior treatment, if they are asymptomatics and without engagement. In cases of symptomatic brain metastases, subjects could be included only if surgery and / or radiotherapy (stereotactic or in toto) were performed and if the cerebral metastatic localization allow IT or intra-ventricular treatment. The last radiotherapy session or the surgery must have been done 3 weeks before.
* Aged 18 years old or more
* Male and female
* Life expectancy more than 2 months
* Satisfactory Cardiac function: left ventricular ejection fraction (LVEF) determined by ultrasound scan or myocardial scintigraphy
* Adequate Biological functions 14 days before inclusion, according to the criteria below: Neutrophils > 1.0 x 109/L, Hemoglobin > 9.0 g/dL (+ transfusion if needed,Platelets > 50 x 109/L,Bilirubin < 3 x N, ALT & AST < 10 x N, Creatinine < 2.0 mg/dL, Clearance > 25 mL/min (Cockcroft and Gault formula), Prothrombin time > 70 %, Kaolin cephalin coagulation time < 1.5 x N.
* Women of childbearing potential, must take adequate birth control measure during the study period and must have a negative pregnancy test (BetaHCG serum)
* The subjects must perform all evaluations of pre-inclusion, as provided by the protocol
* Signed written inform consent

Exclusion Criteria:

* CSF circulation disorders suspected on MRI brain (obstructive hydrocephalus) or medullar (obstacle) with, in case of a focal radiotherapy on obstructive lesion, checking the restoration of transit traffic by isotope CSF
* Anti-coagulant effective dose treatment when trastuzumab administration by lumbar puncture
* Patient on Lapatinib (wash out> 2 weeks from the date of first dose intrathecal trastuzumab)
* Known or suspected trastuzumab allergy
* Contraindications of trastuzumab administration, including cardiac diseases: LVEF <laboratory lower limit of normal or any other heart condition which would expose the subject to an unreasonable risk if he were to participate in the study
* Severe toxicity unresolved or unstable related to another previous study restricted drug and / or a cancer treatment
* Ventriculoperitoneal or atrial shunting excepted if the valve could be turn off (on-off switch) and the patient can stand it during 6 h after each injection of trastuzumab
* Dementia, altered mental status or psychiatric condition that would prevent the subject to understand or give informed consent
* Pre-existing severe cerebrovascular disease, such as stroke in a major vessel, vasculitis in the central nervous system or malignant hypertension
* Uncontrolled infection
* Participation in a clinical study with an experimental molecule
* No affiliation to a Social insurance (beneficiary or assignee)
* Pregnant women, breastfeeding or of childbearing age not taking contraceptive
* Subject unable to make follow up schedule
* Persons deprived of liberty or under guardianship (including curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Phase I : To determine the Trastuzumab maximum tolerated dose (MTD) when weekly administrated by intrathecal or intraventricular route. | 2 months
  Phase I : To determine the Trastuzumab maximimum tolerated dose (MTD) when weekly administrated by intrathecal or intraventricular route to reach a intra CSF target concentration (30 µg/mL) near the conventional therapeutic concentration and depending on the dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Phase I : Recommended dose (RD will be used in Phase II) | 2 months
Phase I&II : Toxicity during treatment | 2 months
  Issued the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 National Cancer Institute (NCI)
Time to neurologic progression | 2 years
Biological response: CSF cellularity and protein concentration | 2 years
Radiological response: cerebrospinal meningitis and neuraxis MRI | 2 years
Impact on quality of life | 2 years
Impact on survival (overall survival, survival without neurological progression, progression-free survival) | 2 years
Pharmacokinetics: dose of trastuzumab in CSF and plasma | 2 months
FCGR3A Genetic status influence on efficacy trastuzumab in metastatic breast cancer | 2 years
Phase II : Determination of antitumor activity trastuzumab when administrated by IT or intra-ventricular in terms of neurological progression free survival at 2 months | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Maya Gutierrez, MD, Study Director — Institut Curie - Hopital Rene Huguenin - Saint-Cloud - France
Locations (10):
- France (10):
  - François Baclesse Center, Caen, Calvados
  - Rene Huguenin Hospital, Saint-Cloud, Haut de Seine
  - Oscar Lambret Center, Lille, Nord
  - Léon Bérard Center, Lyon, Rhone
  - Institut Bergonié, Bordeaux
  - CHU Grenoble, Grenoble
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Univesitaire du Cancer de Toulouse, Toulouse
  - Institut Curie - Claudius Regaud Hospital, Paris, Île-de-France Region
  - Pitie Salpetriere Hospital, Paris, Île-de-France Region

REFERENCES:
- [Result] Bonneau C, Paintaud G, Tredan O, Dubot C, Desvignes C, Dieras V, Taillibert S, Tresca P, Turbiez I, Li J, Passot C, Mefti F, Mouret-Fourme E, Le Rhun E, Gutierrez M. Phase I feasibility study for intrathecal administration of trastuzumab in patients with HER2 positive breast carcinomatous meningitis. Eur J Cancer. 2018 May;95:75-84. doi: 10.1016/j.ejca.2018.02.032. Epub 2018 Apr 7. PMID 29635147